CLINICAL TRIAL: NCT00927914
Title: A 2-year, Randomized, Double-blind, Placebo-controlled, Multi-center, Phase II-III Study to Evaluate the Efficacy and Safety of Oral Ranirestat (40 and 80 mg) in Mild to Moderate Diabetic Sensorimotor Polyneuropathy
Brief Title: Evaluating the Efficacy and Safety of Oral Ranirestat (40 and 80 mg) in Mild to Moderate Diabetic Sensorimotor Polyneuropathy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AS3201-G000-291; 2008-002843-18 (EudraCT Number)
Record Dates: First submitted 2009-06-24; First posted 2009-06-25 (Estimated); Last update posted 2019-02-21 (Actual); Status verified 2015-11

CONDITIONS: Mild to Moderate Diabetic Sensorimotor Polyneuropathy
MeSH Terms: interventions — ranirestat

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Ranirestat 80 mg (Experimental): Two 80 mg Ranirestat tablets, given orally, once daily, preferably in the morning with or without a light breakfast, for upto 24 months.
  Interventions: Drug: Ranirestat
- Ranirestat 40 mg (Experimental): One 40 mg tablet of Ranirestat and a matching placebo, given orally, once daily, preferably in the morning with or without a light breakfast, for upto 24 months.
  Interventions: Drug: Ranirestat; Drug: Placebo
- Placebo (Placebo Comparator): Two placebo tablets, given orally, once daily, preferably in the morning with or without a light breakfast, for upto 24 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ranirestat — Ranirestat 40 mg tablets
  Arms: Ranirestat 40 mg; Ranirestat 80 mg
Drug: Placebo — Placebo tablets
  Arms: Placebo; Ranirestat 40 mg

SUMMARY:
The purpose of this study is to determine the effect of 40 mg and 80 mg ranirestat on peroneal motor nerve conduction velocity relative to placebo in subjects with mild to moderate diabetic sensorimotor polyneuropathy.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with Type 1 or Type 2, insulin-dependent or non insulin-dependent diabetes mellitus.
* Subjects with a history of distal symmetric polyneuropathy, secondary to diabetes, diagnosed in accordance with the American Academy of Neurology criteria.
* Female subjects, who are of non-reproductive potential (>=12 months post-menopausal or surgically sterile) or who are using adequate contraception which includes abstinence or double barrier methods (diaphragm and condom with spermicidal cream, intrauterine device and condom with spermicidal cream). Male subjects with partners of child-bearing potential must also use adequate contraception.
* Subjects must be able to read, understand, and provide written informed consent before enrolling in the study at screening.

Exclusion Criteria:

* History of diabetic foot ulcers or lower extremity amputation.
* Diabetic amyotrophy or non-diabetic cause of lower limb neuropathy/neuropathic symptoms.
* Clinically significant illness which, in the opinion of the investigator, would compromise a subject's suitability to participate in the study for reasons of safety or would confound the efficacy assessments.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Actual)
Dates: Start 2009-07 (Actual); Primary Completion 2013-01 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Peroneal motor nerve conduction velocity: the mean of duplicate bilateral recordings made within 1-21 days of each other. | 24 months

SECONDARY OUTCOMES:
Neuropathy total symptom score-6 via a self-administered questionnaire and vibration perception threshold recorded with a neurothesiometer. | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Roderick Junor, Study Director — Eisai Limited
Locations (1):
- The Johns Hopkins Hospital, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Polydefkis M, Arezzo J, Nash M, Bril V, Shaibani A, Gordon RJ, Bradshaw KL, Junor RW; Ranirestat Study Group. Safety and efficacy of ranirestat in patients with mild-to-moderate diabetic sensorimotor polyneuropathy. J Peripher Nerv Syst. 2015 Dec;20(4):363-71. doi: 10.1111/jns.12138. PMID 26313450